CLINICAL TRIAL: NCT04993352
Title: A Phase I/II, Single-arm, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of HLX04-O Administered by Intravitreal Injection in Subjects With Wet Age Related Macular Degeneration (wAMD)
Brief Title: Evaluate the Safety and Efficacy of HLX04-O in Subjects With wAMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX04-O-wAMD-CN01
Record Dates: First submitted 2021-07-08; First posted 2021-08-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Vascular Endothelial Growth Factor A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX04-O (Experimental): Biologic recombinant anti-VEGF humanized monoclonal antibody.
  Interventions: Drug: recombinant anti-vascular endothelial growth factor (VEGF) humanized monoclonal antibody ophthalmic injection

INTERVENTIONS:
Drug: recombinant anti-vascular endothelial growth factor (VEGF) humanized monoclonal antibody ophthalmic injection — 0.05mL (12.5mg/0.5mL/vial) HLX-04-O solution at a 4-week interval for intravitreal injection

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of HLX04-O administered every 4 weeks in participants with wet age-related macular degeneration (wAMD)

DETAILED DESCRIPTION:
This is a Phase I/II, Single-arm, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of HLX04-O Administered by Intravitreal Injection in Subjects with wet Age related Macular Degeneration (wAMD).The study will be conducted in approximately 6 sites in China.

ELIGIBILITY:
Inclusion Criteria:

1. Capable to fully understand and sign the informed consent form (ICF).
2. Women or men aged ≥50 years when signing the ICF.
3. Newly diagnosed or recurrently, active subfoveal or juxtafoveal CNV lesions secondary to AMD in the study eye. (Active CNV was defined as leakage on FA and subretinal or intraretinal fluid on OCT).
4. The total lesion area (including bleeding, scar and neovascularization) of the study eye ≤12 disc area (DA).
5. The BCVA letters between 15 and 78, inclusive, in the study eye, using Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
6. Clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm the diagnosis.

Exclusion Criteria:

1. Macular-related retinal pigment epithelial tears in the study eye; scar, fibrosis or atrophy involving the fovea, or CNV due to other causes in the study eye (e.g., ocular histoplasmosis, trauma, or pathological myopia, etc.).
2. The fellow (non-study) eye needs anti-VEGF IVT injection (e.g. CNV due to wAMD, trauma, pathological myopia, retina vein occlusion, diabetic macular edema, etc) in the next 3 months, in the investigator's judgment.
3. Active or recent (within 1 month prior to dose 1) intraocular, extraocular or periocular infection (including but not limited to conjunctivitis, keratitis, scleritis or endophthalmitis), or history of idiopathic or autoimmune-associated uveitis in either eye.
4. Vitreous hemorrhage in study eye within 3 months prior to dose 1.
5. Aphakia (except intraocular lens) or posterior capsular rupture of the lens (except yttrium aluminium-garnet (YAG) laser posterior capsulotomy after intraocular lens implantation ≥1 month prior to first dose) in the study eye.
6. Corneal dystrophy or history of corneal transplantation, scleral softening or history of scleral softening, history of rhegmatogenous retinal detachment or macular hole (Stage II, III or IV) in the study eye.
7. Uncontrolled glaucoma (defined as intraocular pressure [IOP] ≥25 mmHg despite treatment with antiglaucoma medication), and/or glaucoma filtering surgery (e.g., trabeculectomy, scleral nipping, non-penetrating trabeculectomy, etc.).
8. Equivalent spherical diopter of the study eye ≥-8D. For participants who had undergone refractive correction or cataract surgery, the equivalent spherical diopter of the study eye before surgery ≥-8D.
9. Estimated by the Investigator, any concurrent intraocular condition except wAMD (e.g., diabetic retinopathy, dry AMD, retina vein occlusion, uveitis, angioid streaks, retinal detachment, macular epiretinal membrane, amblyopia, central serous chorioretinopathy, etc.) in the study eye that limited the potential to gain visual acuity upon treatment with the investigational product, or could have required medical or surgical intervention during the study to prevent or treat visual loss.
10. Underwent intraocular surgery including verteporfin photodynamic therapy (PDT), transpupillary thermotherapy, macular translocation, vitrectomy, laser photocoagulation in macular area, other surgery in macular area or surgery to treat AMD.
11. Previous intraocular or periocular surgery within 1 month prior to dose 1(including laser photocoagulation in juxtafoveal, cataract surgery, etc.), or current unhealed wound, moderate or severe ulcer or history of fracture in the study eye.
12. Subconjunctival or intraocular or systemic use of corticosteroids within 3 months (including subconjunctival or intraocular long-acting implant within 6 months).
13. Previous systemic anti-VEGF therapy or IVT injection of any anti-VEGF drug into either eye or other ocular use of anti-VEGF drug (ranibizumab, aflibercept or conbercept) within 3 months prior to dose 1.
14. Participated in any drug (other than vitamins and minerals) or device clinical trials within 3 months or the duration of 5 half-lives of the study drug (which is longer) prior to dose 1 and have used the test drug or received device treatment.
15. Pregnancy or lactation.
16. Men or women fail to meet both of the following ones: 1) women must have a negative serum pregnancy test result within 14 days prior to initiation of the study intervention; 2) agreement to remain abstinent (refrain from heterosexual intercourse) or use effective contraceptive methods from signed ICF to at least 6 months following the last dose of the study intervention. Effective contraceptive methods include bilateral tubal ligation, male sterilization, established physical contraception and copper intrauterine devices (IUDs).
17. Stroke or myocardial infarction within 6 months prior to dose 1, uncontrolled hypertension (systolic blood pressure≥160 mmHg, or diastolic blood pressure ≥100 mmHg), etc.
18. Uncontrolled diabetes (defined as HbA1c>10.0%).
19. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) is more than twice the upper limit of normal (ULN), and/or serum creatinine is 1.2 times more than the ULN, and is clinically significant in the opinion of the Investigator.
20. Abnormal coagulation function（prothrombin time ≥ 3 seconds over ULN, activated partial thromboplastin time ≥ 10 seconds over ULN）
21. Active disseminated intravascular coagulation and obvious bleeding tendency within 3 months prior to dose 1.
22. Evidence of significant uncontrolled concomitant diseases such as cardiovascular diseases, nervous system diseases, respiratory system diseases, urinary system diseases, digestive system diseases and endocrine diseases.
23. Current treatment for active systemic infection, or history of recurrent serious infections.
24. Known active or suspected autoimmune diseases, requiring systemic immunosuppressive therapy.
25. Positive for syphilis screening test or positive for human immunodeficiency virus (HIV) screening test.
26. Known allergy to any component of the study intervention or history of allergy to fluorescein(only for patients who cannot undergo OCT-A examination but have to undergo ICGA examination) or indocyanine green, any anesthetics or antimicrobial agents used during the course of the study.
27. Participant who has been diagnosed to be COVID-19 within 1 month prior to dose 1 or who has received COVID-19 vaccine within 1week prior to dose 1.
28. In the Investigator's judgment, there is evidence of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the participant at high risk for treatment complications, or other conditions considered not amenable to this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Phase I: Safety events | week 4
  toxicity and causality (related to or possibly related to HLX04 O) that occurs within 4 weeks after the first treatment (single administration)
Phase 2: Mean change of letters from baseline in the BCVA at Week 12 | Week 12
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

SECONDARY OUTCOMES:
Phase I: HLX04-O systemic PK parameters following IVT administration of Dose 1 and Dose 4 | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: Mean change of letters from baseline in the BCVA over time | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: Proportion of patients gaining at least 15/10/5 letters in the BCVA at Week 12, 24, 36 and 48 | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: Mean change from baseline in the total area of CNV and the total area of fluorescein leakage on fluorescein angiography (FA) at Week 12, 24 and 48 | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: Mean change from baseline in central retina thickness (CRT) on optical coherence tomography (OCT) at Week 12, 24, 36 and 48 | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: Change from baseline in NEI VFQ-25 scale score at Week 12, 24, and 48 | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: Percentage and severity of ocular AEs (IVT procedure related and Investigation Medication related), non-ocular AEs; laboratory abnormalities; vital sign, physical examination abnormalities, etc. | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: Incidence of ADAs and NAbs against HLX04-O following IVT administration | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Phase 2: • HLX04-O serum concentrations before Dose 1, 168 hours after Dose 1, before Dose 2, before Dose 4, 168 hours after Dose 4, before Dose 5, before Dose 8, before Dose 12 and the last visit | 1 year
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

CONTACTS AND LOCATIONS:
Locations (1):
- XuZhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Wu Y, Lyu YL, Chang MQ, Xu QJ, Liu YM, Kang WY, Wang QY, Li CL. Efficacy and safety of intravitreal HLX04-O, an anti-VEGF monoclonal antibody, for the treatment of wet age-related macular degeneration. Int J Ophthalmol. 2022 Sep 18;15(9):1549-1553. doi: 10.18240/ijo.2022.09.20. eCollection 2022. PMID 36124180